CLINICAL TRIAL: NCT05022485
Title: Performance, Safety and Clinical Benefits of a Noble Metal Alloy-coated Intramedullary Nail: a Multicenter, Prospective Trial With a Retrospective Control
Brief Title: Zimmer® Natural Nail® (ZNN) Bactiguard Tibia Post-Market Clinical Follow-up Study
Status: Recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CMG2020-32T
Record Dates: First submitted 2021-07-16; First posted 2021-08-26 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Tibial Fractures; Fracture Infection
Keywords: intramedullary tibia nail; Bactiguard
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Investigational group: Subjects that will be implanted with the ZNN Bactiguard tibia device.
  Interventions: Device: ZNN Bactiguard tibia
- Control group: Subjects that have received an uncoated titanium-alloy tibia nail in the past (data collection is retrospective; patients will not have to undergo any study-related procedure).

INTERVENTIONS:
Device: ZNN Bactiguard tibia — Tibia fracture fixation
  Groups: Investigational group

SUMMARY:
Primary objective of this study is to compare fracture related infection (FRI) rates of ZNN Bactiguard Tibia to conventional uncoated titanium-alloy nails 12 months after tibia fracture fixation.

The secondary objectives are confirmation of safety, performance and clinical benefits of ZNN Bactiguard implant and related instrumentation12 months after fracture fixation.

DETAILED DESCRIPTION:
This is a multicenter, prospective, Post-market Clinical Follow-up (PMCF) Study with retrospective controls.

The study will enroll patients that will be implanted with the Zimmer Natural Nail Bactiguard Tibia device and retrospective controls implanted with standard titanium-alloy tibia nails.

500 tibias will be recruited at maximum 15 sites and allocated on a 1:1 ratio into an:

* investigational group (prospective/consecutive series of 250 tibias treated with ZNN Bactiguard tibia)
* a control group (retrospective series of 250 tibias treated with uncoated titanium-alloy tibia nail - data collection will be retrospective, these subjects will not have to undergo any study-related procedure).

The primary endpoint is the Fracture Related Infection (FRI) rate in the study population 12 months after fracture fixation.

The secondary endpoint is the confirmation of safety, performance and clinical benefits of ZNN Bactiguard implant and related instrumentation through the following measure systems:

* Radiologic (RUST) & clinical (FIX-IT) fracture healing 12 months after fracture fixation (performance).
* Patients' outcomes assessed by the Oxford Knee Score 12 months after fracture fixation (clinical benefits).
* EQ5D-5L (patients' quality of life).
* Incidence and frequency of adverse events (safety).

Data will be collected at 2 weeks, 3 months, 6 months and 1 year after fracture fixation.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 or older.
* Patient has signed IRB/EC-approved informed consent (if applicable for retrospective controls, based on local requirements).
* Patient suffered primary tibia fracture (monolateral or bilateral) at high risk of infection, eligible for fixation by intramedullary (IM) nailing (standard or suprapatellar approach) and meets at least one of the following conditions:

  * Open fractures (incl. gunshot fractures): Gustilo Type I, II, III A and III B.
  * Delayed treatment (initial treatment by external fixation due to swelling/ high energy trauma followed by definitive treatment by intramedullary nail).
  * Fracture associated with ipsilateral leg compartment syndrome treated with fasciotomy wound(s).
  * Closed fractures with severe tissue damage: Tscherne grade C2 and C3.
* Patient:

  * will be treated with ZNN Bactiguard tibia for inclusion in investigational group (retrospective enrollment is allowed up to 1st follow-up visit);
  * was treated with uncoated (conventional) titanium-alloy intramedullary tibia nail for inclusion in control group;

Exclusion Criteria:

* Patient is unwilling or unable to give consent.
* Patient is not expected to survive follow-up schedule.
* Patient is anticipated to be non-compliant to the study protocol.
* Patient has a mental or neurological condition or alcohol/drug addiction that will not allow for proper informed consent and/or participation in follow-up program.
* Patient is a prisoner.
* Patient is known to be pregnant and/or breastfeeding.
* Patient suffered tibia fracture that meets any of the following conditions:

  * Pathologic fracture.
  * Gustilo Type IIIC open fracture.
  * Patient has multisegmented fracture NOT eligible for fixation by intramedullary nailing.
  * Patients with wound closure more than 10 days after injury.
  * Besides IM nail, patient requires additional tibia fixation by plate (additional tibia fixation by screw(s) and/or fibula plate fixation are allowed).
  * Concomitant with fracture, patient suffered head injury with Abbreviated Injury Score (AIS) ≥ 3.
* For control group:

  * patient doesn't have all the minimum required data available:

    1. demographic information
    2. injury classification
    3. FRI information
    4. operative report and device information
    5. radiographic analyses (until fracture healing or confirmation of non-union leading to reoperation)
* Tibia medullary canal is obliterated by a previous fracture or tumor*
* Tibia bone shaft having excessive bow or a deformity*
* Lack of bone substance or bone quality, which makes stable seating of the nail implant impossible*
* All concomitant diseases that can impair the operation, functioning or the success of the nail implant*
* Insufficient blood circulation*
* Skeletally immature patients*
* Infection*

  * ZNN Bactiguard tibia contraindication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18-year-old patients or older with tibia fractures at high risk for infection (as defined in the inclusion criteria) treated with a titanium-alloy intramedullary nail.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Fracture related infection (FRI) rate in investigational and control group | 12 months after fracture fixation
  FRI diagnosed according to the updated diagnostic algorithm drafted by the Fracture-Related Infection Consensus Group (Definition and diagnosis of fracture-related infection, M McNally,G Govaert, M Dudareva, M Morgenstern, W J Metsemakers, EFORT Open Rev 2020;5:614-619.)

SECONDARY OUTCOMES:
Tibia fracture healing assessed radiologically through Radiographic Union Scale in Tibial fractures (RUST) score | 12 months after fracture fixation
  The RUST score assigns each tibial cortex (anterior, posterior, medial and lateral) a score from 1 to 3, based on the appearance on the X-ray. The scores of all cortices combined will give a minimum score of 4 (definitely not healed) up to a maximum of 12 (completely healed).
Tibia fracture healing assessed clinically through the Function IndeX for Trauma (FIX-IT) score | 12 months after fracture fixation
  The FIX-IT score assesses the subject's pain and ability to bear weight on lower extremity fractures. It ranges from 0 to 12 points, with 12 points representing the highest level of limb function.
Limb functionality measured through the Oxford Knee Score | 12 months after fracture fixation
  The Oxford Knee Score consists of twelve questions regarding knee functionality and pain. The score ranges from 12 to 60 points, with 12 points indicating the best outcome.
Quality of life of study participants assessed through the EQ-5D-5L questionnaire | 12 months after fracture fixation
  The EQ-5D is a self-reported descriptive questionnaire about the patient's quality of life composed of 5 questions referring to mobility, self-care, daily activities, pain and anxiety/depression. Each question has 3 possible answers, which define the level of perceived problems (none, moderate,extreme problem)
Incidence and frequency of adverse events | 12 months after fracture fixation
  Frequency and incidence of recorded AEs will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Rohmer, Study Director — Clin Ops Director
Locations (16):
- Tirolkliniken Innsbruck, Innsbruck, Austria
- France (2):
  - Hôpital Ambroise-Paré, Boulogne-Billancourt
  - Hôpitaux Universitaires de Marseille Nord, Marseille
- Germany (3):
  - Universitätsklinikum Marburg, Marburg, Hesse
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsklinikum Regensburg, Regensburg
- Italy (2):
  - AOU Policlinico di Bari, Bari
  - Azienda Ospedaliero-Universitaria Careggi, Florence
- South Africa (2):
  - Tygerberg Hospital, Cape Town
  - Groote Schuur Hospital, Cape Town
- Hospital Universitario Valle de Hebrón, Barcelona, Catalonia, Spain
- Kantonsspital Winterthur, Winterthur, Canton of Zurich, Switzerland
- United Kingdom (4):
  - Royal Infirmary of Edinburgh, Edinburgh
  - Leeds General Infirmary, Leeds
  - The Royal London Hospital, London
  - King's College Hospital NHS Trust, London